CLINICAL TRIAL: NCT03875924
Title: Multicenter Retrospective Study From 5 Hemostasis Treatment Centers in Western France: Severe Hemorrhagic Treated Occurrences' Patterns and Global Substitutive COagulation Factors THerapy in the Inherited Von WILLebrand Disease
Brief Title: REAL-LIFE DATA OF CONSTITUTIONAL VON WILLEBRAND DISEASE IN WESTERN FRANCE (HOPSCOTcH-WILL)
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: CHU de Brest (Unknown); University Hospital, Angers (Other Government); CH Le Mans (Unknown); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0075
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VWD BERHLINGO: Patients with constitutional von Willebrand Disease, of any severity, with or without inhibitor followed in one of the investigator centers
  Interventions: Other: VWD treatments

INTERVENTIONS:
Other: VWD treatments — Modalities and types of treatments in VWD patients for severe hemorrhagic events: INN, quantities, duration of treatment

SUMMARY:
Von Willebrand disease (VWD) is the most common constitutional bleeding disorder in the world, caused by missing or defective von Willebrand factor (VWF). In France, VWD affects approximatively 7,000 patients.

There are many types of VWD. The severest forms are characterized by the occurrence of extremely serious bleedings, requiring in-stays with clotting factors (CF) treatments in specialized hospital units and/or an ambulatory substitutive therapy; both of them are highly expensive.

In France, Hemostasis Treatment Centers (HTC) have the opportunity to record these kinds of data in a database called NHEMO (Net-Hemostasis = care database for constitutional bleeding disorders). Further ahead, the data can be coded, dumped into and extracted from the research database BERHLINGO and analyzed.

The HOPSCOTcH-WILL study will be a retrospective, non-interventional, multicenter (national) cohort study & will provide an overview of the real-life management of patients with VWD in western France requiring a substitutive treatment with VWF, as well as a description of the characteristics of their hemorrhagic events.

Model : Observationnal, real world evidence study. Time Horizon : 2015-2018. HTC (France): Western University Hospitals (BERHLINGO network) = Nantes University Hospital (promotion), Angers University Hospital, Brest University Hospital, Le Mans Regional Hospital & Rennes University Hospital

DETAILED DESCRIPTION:
von Willebrand Disease (vWD) represents the most common autosomal inherited bleeding disorders with a prevalence up to 1%; nevertheless the clinical relevant patients represent only 0.01% of the population.

vWD is caused by a deficiency and/or abnormality of von Willebrand factor (VWF), inhibiting a satisfactory hemostasis. vWD is usually classified into three main types according to quantitative (Types 1 and 3) or qualitative (Types 2A, 2B, 2M, 2N) deficiencies. Type 3 patients have the highest bleeding risk, type 2 patients are intermediate and type 1 patients have the lowest bleeding risk. Beyond the typology, VWF levels, and therefore the hemorrhagic exposition, are also notably influenced by physiological (age, exercise, pregnancy, gene mutations) or pathological (inflammation and cancer) variables. Furthermore, blood group plays a major role in plasma VWF levels; in fact they are 25%-35% lower in type-0 individuals than in non-0. As a result, the clinical and biological identification of vWD can be extremely challenging and may lead to a delay in the diagnosis.

In vWD, the clinical manifestations are essentially mucosal bleeding symptoms. Epistaxis, menorrhagia, easy bruising, gingival bleeding are flagrant manifestations of the disease and, despite the mostly small somatic impact in the majority of patients; they may significantly affect the quality of life. Nevertheless, severe affected patients may face upper consequences: gastrointestinal (GI) bleeding may be particularly frequent and difficult to manage, and they are as well at high risk to develop major and life-threatening bleeds after surgical procedures, even after minor ones such as tooth extraction.

To guarantee the best medical care management, VWD patients are followed in specialized rare disease centers, both for the ambulatory follow-up and the hospitalizations & outpatient aftercare. These hospital structures are the only ones authorized to prescribe and dispense in- & outpatients' substitutive treatments.

Indeed, the optimal effective treatment of the disorder is the replacement of VWF by using VWF concentrate obtained by fractionation of human plasma; in emergency, recombinant or plasma-derived factor VIII (FVIII) can be added to the VWF. In case of history of inhibitors, high dose of FVIII or by-passing agents can also be used. The current treatment for vWD involves intravenous injections of VWF that are either given on demand in response to a bleeding event or as a prophylactic therapy that is administered 2 to 4 times a week. Numerous studies have shown the efficacy of prophylactic therapy in severe patients, but the investigators lack data about surgery procedures and perioperative management. Moreover, regardless of the small amounts of patients, those treatments remain quite costly and may represent an economic burden for the Assurance Health System.

Due to the future availability of the first recombinant VWF, the investigators need a better understanding of the current French practices. The lack of literature on the topic is undeniably blatant and the few relevant papers concerned specific pd-VWF concentrates; no RWD publication has been identified for the specific French cohort. The heterogeneity of VWD concentrates brands and VWD types make the development of personalized care quite difficult in this context and more information is needed, especially for the peri-operative treatment. The economic evaluations usually focus on prophylaxis treatments or a specific concentrate, neglecting a significant percentage of patients.

The objective of our 4-years retrospective study HOPSCOTcH-WILL is to provide an accurate and detailed account of current vWD therapeutic management by collecting real-life data on hemorrhagic treated events in 5 Western French HTC (Angers, Brest, Le Mans, Nantes & Rennes). The data will be retrospectively recorded during 48 months from 2015 to 2018 for patients followed in the 5 HTC involved in the study. A focus will be done on GI episodes and surgeries which are the most at risk hemorrhagic events in vWD.

HOPSCOTcH-WILL could be considered as reliable photography of Western French HTC at a particular time. Therefore, and especially with the launch of a new recombinant VWF, it is particularly important to get a clear state-of-the-art and to assess the economic impact for the French Health System.

ELIGIBILITY:
Inclusion Criteria:

* Constitutional VWD patient, of any severity, with or without inhibitors (according to the CRMW criteria*),
* Patient included in the research database BERHLINGO
* Patient treated or not by desmopressin or VWF/FVIII/by-passing agents available on the French market (at baseline)
* Patient who agrees to participate in the HOPSCOTcH and followed in one of the 5 investigator HTC
* Patient who are not under guardianship

  * CRMW criteria for constitutional VWD definition:

Severe forms: VWF:Ag and VWF:RCo <5 UI/dL VWD 2A or 2M: VWF:RCo/VWF:Ag < 0.7 and/or ratio VWF:CB/VWF:Ag < 0.7 VWD 2B: unexplained thrombopenia and/or positive RIPA < 0.8 mg/mL (for any value of VWF:RCo/VWF:Ag) VWD 2N: FVIII:C/VWF:Ag < 0.6 and reduced to very reduced VWF:FVIIIB VWF:Ag <30 UI/dL (in the absence of every previous criteria)

Exclusion Criteria:

* Patients Under guardianship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: On 16th July 2018, 919 constitutional VWD* patients are included in the NHEMO database for the 5 Western France BERHLINGO HTC = Angers, Brest, Le Mans, Nantes & Rennes. In case of hemorrhagic events:
  * 16.4% (n=151) are likely to be treated with desmopressin only,
  * 20.8% (n=191) with CF only - i.e. von Willebrand Factor (VWF) and/or Factor VIII (FVIII) and /or by-passing agents -,
  * 21.6% (n=199) with desmopressin and/or CF. To be taken into account: 41.2% of patients have no treatment mentioned or are in a phase of evaluation of their modalities of treatment (=desmopressin test to be done or desmopressin treatment to be debated before use, essentially).
  It is estimated that out of these potential treated patients, 300 could have been treated with CF at least once during the 4-years period.
  *According to the CRMW criteria for constitutional VWD
Sampling Method: Non-Probability Sample
Enrollment: 926 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients of any severity (in and outpatients care consumptions) | Every treatment over 48 months

SECONDARY OUTCOMES:
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, by type of VWD (in and outpatients care consumptions) | Every treatment over 48 months
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, according the history of inhibitor (in and outpatients care consumptions) | Every treatment over 48 months
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, by regimen of treatment (in and outpatients care consumptions) | Every treatment over 48 months
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, by type of treatment (pdVWF, FVIII, pdVWF/FVIII, desmopressin) | Every treatment over 48 months
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, by type of hemorrhage | Every treatment over 48 months
Consumptions of clotting factors/desmopressine for the treatment of severe hemorrhagic events in VWD patients, by age and sex | Every treatment over 48 months
Cost of illness study from the French payer perspective for the von Willebrand Disease | Over 48 months
Estimation of the annual treated bleeding rate (ABR) in VWD patients | Over 48 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Le Mans Regional Hospital, Le Mans
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horvais V, Beurrier P, Cussac V, Pan-Petesch B, Schirr-Bonnans S, Rose J, Bayart S, Ternisien C, Fouassier M, Sigaud M, Babuty A, Drillaud N, Guillet B, Trossaert M; BERHLINGO Consortium. Key Drivers of Coagulation Factor Use in Von Willebrand Disease During Hospitalization: An Overview of the French BERHLINGO Cohort. Clin Drug Investig. 2024 Jan;44(1):35-49. doi: 10.1007/s40261-023-01323-1. Epub 2023 Nov 30. PMID 38036930